CLINICAL TRIAL: NCT03483025
Title: Prospective Single Center Randomized Double Blind Controlled Tolerability Trial of Six Hair Cleansing Conditioners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: A17-335
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-04

CONDITIONS: Irritant Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Irritant

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The six hair cleansing products will be packaged in identical 1 ml capped tuberculin syringes (with no needles) and provided to participants. Each syringe will be labeled with the forearm location for application. Identical syringes containing the six hair cleansing products will be dispensed. Treatment site allocation will be determined by a computer-generated randomization log.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Hair Cleansing product 1 (Other): Skin Testing of Hair cleansing products all pts will test 6 hair cleansing products, but site of testing will be randomized and blinded
  Interventions: Other: Skin Testing of Hair cleansing products
- Hair cleansing product 2 (Other): Skin Testing of Hair cleansing products all pts will test 6 hair cleansing products, but site of testing will be randomized and blinded
  Interventions: Other: Skin Testing of Hair cleansing products
- Hair cleansing product 3 (Other): Skin Testing of Hair cleansing products all pts will test 6 hair cleansing products, but site of testing will be randomized and blinded
  Interventions: Other: Skin Testing of Hair cleansing products
- Hair cleansing product 4 (Other): Skin Testing of Hair cleansing products all pts will test 6 hair cleansing products, but site of testing will be randomized and blinded
  Interventions: Other: Skin Testing of Hair cleansing products
- Hair cleansing product 5 (Other): Skin Testing of Hair cleansing products all pts will test 6 hair cleansing products, but site of testing will be randomized and blinded
  Interventions: Other: Skin Testing of Hair cleansing products
- Hair cleansing product 6 (Other): Skin Testing of Hair cleansing products all pts will test 6 hair cleansing products, but site of testing will be randomized and blinded
  Interventions: Other: Skin Testing of Hair cleansing products

INTERVENTIONS:
Other: Skin Testing of Hair cleansing products — 6 different commercially available shampoos

SUMMARY:
Hair cleansing product tolerability study

DETAILED DESCRIPTION:
Study Aim: The objective of this study is to evaluate the tolerability of daily use of f hair cleansing products.

Background/Study Rational/Significance: There have been consumer reports of irritancy and hair loss with use of Wen cleansing conditioner. A recent study of 142 patients found no increase in hair loss when used in normal subjects, however skin assessments for tolerability were not evaluated.

Methodology: This double-blind, randomized, controlled clinical trial will evaluate the tolerability of six hair cleansing products including Wen cleansing conditioner using two standard clinical and research methods, Repeat Open Application Tests (ROAT) (a test for irritancy) and Semi-Open Patch Tests (a test for allergenicity). For the ROAT, participants will apply the hair cleansing products to 6 separate locations on the forearm using a standardized, protocol and scored using a 10-point scale. Application site of each cleansing product will be randomized. Exposure time will be increased in a step-wise fashion over 5 weeks. Participants and investigators will be blinded to location of products. The primary outcome is intolerance; intolerance will be defined as 1) ROAT skin component scoring >6 (of 10 maximum) or 2) ROAT global score of >4 (of 5 maximum). If intolerance to a specific product is reached, the ROAT for that product will be discontinued. . Clinical assessments (global scoring and component scoring) will be performed at 0, 2, and 4 and 5 weeks. Primary outcomes will be measured at 5 weeks. Allergenicity is a secondary outcome and will be assessed with semi-open patch tests to the 6 hair cleansing products performed at week 4 and read at week 5

Setting/ patients: Single center study of 200 patients. To represent a broad spectrum of skin barrier function, recruitment will target enrollment of 150 individuals with a no history of childhood eczema (non-atopic) and 50 individuals with a history of childhood eczema (atopic).

Population: Men and women over the age of 18 years old.

ELIGIBILITY:
Inclusion Criteria:• Age of 18 years or older

* Signed and witnessed written informed consent
* Willingness and ability to comply with the study protocol
* For women of child-bearing potential, negative urine pregnancy test at enrollment

Exclusion Criteria:

* The presence of an overt bacterial, viral or fungal infection of the arms
* The presence of any skin condition on the arms that, in the opinion of the investigator, could interfere with study assessments.
* History of bullous skin disorders, psoriasis, ichthyosis, and/or any other chronic skin condition which could result in skin barrier dysfunction (other than atopic dermatitis).
* Treatment with systemic immunosuppressive drugs within 2 weeks of enrollment.
* Treatment with topical antibacterial, antimycotic, or immunosuppressive medications (including topical corticosteroids) on the forearms within 2 weeks of enrollment.
* Use of over-the-counter moisturizers to the forearms in the 3 days prior to protocol commencement.
* Menstruating females of childbearing potential who are not willing to use a medically accepted method of contraception, during the study and up to 4 weeks after the end of study. Medically approved contraception may, at the discretion of the investigator, include abstinence.
* Women who are breastfeeding
* Patients with a severe medical condition(s) which, in the view of the investigator, prohibits participation in the study
* Use of any other investigational agent in the 30 days prior to study commencement
* Known allergy to the study products or ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Repeat Open Application Test | 5 wks
  intolerance will be defined as 1) ROAT skin component scoring >6 (of 10 maximum) or 2) ROAT global score of >4 (of 5 maximum).

CONTACTS AND LOCATIONS:
Overall Officials: erin warshaw, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Park Nicollet Contact Dermatitis Clinic, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warshaw EM, Schlarbaum JP, Liou YL, Kimyon RS, Zhang AJ, Nikle AB, Monnot AD, Hylwa SA. Tolerability of hair cleansing conditioners: a double-blind randomized, controlled trial designed to evaluate consumer complaints to the U.S. Food and Drug Administration. Cutan Ocul Toxicol. 2020 Jun;39(2):89-96. doi: 10.1080/15569527.2020.1722154. Epub 2020 Mar 2. PMID 32122177